CLINICAL TRIAL: NCT02574117
Title: Corticotomy-assisted Slow Maxillary Expansion With Bone Allograft Assessed With Cone Beam Computed Tomography in Young Adults
Brief Title: Cone Beam Computed Tomography for Evaluating Corticotomy-assisted Maxillary Expansion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha Ayman Ghallab, Associate Professor of Oral Medicine and Periodontology, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Corticotomy_CBCT
Record Dates: First submitted 2015-10-08; First posted 2015-10-12 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Posterior Cross Bite
MeSH Terms: interventions — Surgical Flaps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- flap with corticotomy and bone allograft (Experimental): Maxillary expansion with quad helix appliance was applied to posterior teeth with cross bite. Then corticotomy surgical procedure associated with addition of commercially available bone allograft; demineralized freeze-dried bone allograft on the buccal surface of maxillary 1st premolar, 2nd premolar and 1st molar areas.
  Interventions: Procedure: flap with corticotomy and bone allograft

INTERVENTIONS:
Procedure: flap with corticotomy and bone allograft — A maxillary expansion with quad helix appliance was placed on the posterior teeth with cross bite. A Luebke buccal flap was opened in the area of maxillary 1st premolar, 2nd premolar and first molar with a no. 15 scalpel. Corticotomy procedure was performed using low speed round bur size 3, holes to create a 0.5 mm deep hole penetrating the cortical bone. Multiple holes were performed leaving 1.5 mm distance in between. The defects were covered with demineralized freeze-dried bone allograft and the flap was sutured in its original position with 3-0 black silk suture.
  Other Names: periodontally accelerated orthodontics and DFDBA

SUMMARY:
Maxillary expansion was performed for adult female patients suffering from maxillary constriction with bilateral posterior cross-bite using fixed Quad-helix appliance, for about 8 months. The appliance was delivered and activated at the day of corticotomy and bone graft. The activation was made half-molar unit each side. The patient was scheduled each month to activate the appliance or reactivate if needed. Corticotomy was performed at area of maxillary 1st premolar, 2nd premolar and first molar. Cone beam computed tomography was performed, before appliance activation and corticotomy, at the end of expansion (8 months) and after finishing orthodontic treatment (average 2.5 years from start of treatment).

DETAILED DESCRIPTION:
Maxillary expansion was performed for adult female patients suffering from maxillary constriction with bilateral posterior cross-bite & dental arch discrepancy average 12 mm using fixed Quad-helix appliance, for about 8 months. The appliance was delivered and activated at the day of corticotomy and bone graft (demineralized freeze-dried bone allograft). The activation was made half-molar unit each side. The patient was scheduled each month to activate the appliance or reactivate if needed. Corticotomy was performed at area of maxillary 1st premolar, 2nd premolar and first molar. Cone beam computed tomography was performed at three stages.

T1 (baseline) Before appliance activation and corticotomy. T2 At the end of expansion. (about 8 months of expansion). T3 At the finishing stage of orthodontic treatment (average 2.5 years from start of treatment).

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients (18-22 years) suffering from maxillary constriction with bilateral posterior cross-bite.
* Dental arch discrepancy average 12 mm.

Exclusion Criteria:

* Having any given systemic disease.
* Taking any type of medication and/or antibiotic therapy during the 3 months before the study.
* Didn't perform previous orthodontic treatment.
* Current or former smokers.

Ages: 18 Years to 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2010-04; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Inter-arch distance | Change in mm from baseline before surgical procedure to first follow up at 8 months. Change in mm from first follow up at 8 months to second follow up after 2.5 years. Change in mm from baseline to second follow up after 2.5 years.
  Change in mm inter arch distance from baseline before appliance activation and corticotomy till first follow up 8 months after expansion.
  Change in mm inter-arch distance from first follow up 8 months after expansion till second follow up 2.5 years from start of treatment after finishing orthodontic treatment.
  Change in mm inter-arch distance from baseline before appliance activation and corticotomy till second follow up 2.5 years from start of treatment after finishing orthodontic treatment.

SECONDARY OUTCOMES:
Change in tipping angle. | Change from baseline before surgical procedure to first follow up at 8 months. Change from first follow up at 8 months to second follow up after 2.5 years. Change from baseline to second follow up after 2.5 years.
  Change in tipping angle from baseline before appliance activation and corticotomy till first follow up 8 months after expansion.
  Change in tipping angle from first follow up 8 months after expansion till second follow up 2.5 years from start of treatment after finishing orthodontic treatment.
  Change in tipping angle from baseline before appliance activation and corticotomy till second follow up 2.5 years from start of treatment after finishing orthodontic treatment.
Degree of cross bite assessed by measuring mm distance between buccal cusp of the tooth in the upper arch and buccal cusp of same tooth in lower arch. | Change from baseline before surgical procedure to first follow up at 8 months. Change from first follow up at 8 months to second follow up after 2.5 years. Change from baseline to second follow up after 2.5 years.
  Change in degree of cross bite from baseline before appliance activation and corticotomy till first follow up 8 months after expansion.
  Change in degree of cross bite from first follow up 8 months after expansion till second follow up 2.5 years from start of treatment after finishing orthodontic treatment.
  Change in degree of cross bite from baseline before appliance activation and corticotomy till second follow up 2.5 years from start of treatment after finishing orthodontic treatment.
Dehiscence score. | Assessment of the score at First follow up at 8 months and at Second follow up after 2.5 years.
  Dehiscence is the amount of buccal alveolar bone loss around the root surface.
  Dehiscence score as follows; score 0: No Dehiscence. score 1: Dehiscence in cervical third of root only. score 2: Dehiscence in cervical third and middle third of root surface only. score 3: Dehiscence in cervical third and middle third and apical third of root surface.
  Dehiscence is assessed at first follow up 8 months after expansion and at the second follow up 2.5 years from start of treatment after finishing orthodontic treatment.
Buccal bone thickness. | First follow up at 8 months. Second follow up after 2.5 years.
  Assessment of the Buccal bone thickness at first follow up 8 months after expansion and at second follow up 2.5 years from start of treatment after finishing orthodontic treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Khalifa, MD, Principal Investigator — Associate Professor of Oral and Maxillofacial radiology, Faculty of Oral and Dental Medicine, Cairo University.; Eman Mohii, MD, Principal Investigator — Lecturer of Orthodontics, Faculty of Oral and Dental Medicine, Cairo University.; Noha Ghallab, MD, Principal Investigator — Associate Professor of Oral Medicine and Periodontology, Faculty of Oral and Dental Medicine, Cairo University.
Locations (1):
- Faculty of Oral and Dental Medicine, Cairo University, Cairo, Egypt

REFERENCES:
- [Background] Cano J, Campo J, Bonilla E, Colmenero C. Corticotomy-assisted orthodontics. J Clin Exp Dent. 2012 Feb 1;4(1):e54-9. doi: 10.4317/jced.50642. eCollection 2012 Feb. PMID 24558526
- [Background] Shoreibah EA, Ibrahim SA, Attia MS, Diab MM. Clinical and radiographic evaluation of bone grafting in corticotomy-facilitated orthodontics in adults. J Int Acad Periodontol. 2012 Oct;14(4):105-13. PMID 23210199
- [Background] Shoreibah EA, Salama AE, Attia MS, Abu-Seida SM. Corticotomy-facilitated orthodontics in adults using a further modified technique. J Int Acad Periodontol. 2012 Oct;14(4):97-104. PMID 23210198
- [Background] Kim SH, Kim I, Jeong DM, Chung KR, Zadeh H. Corticotomy-assisted decompensation for augmentation of the mandibular anterior ridge. Am J Orthod Dentofacial Orthop. 2011 Nov;140(5):720-31. doi: 10.1016/j.ajodo.2009.12.040. PMID 22051493
- [Background] Hassan AH, Al-Saeed SH, Al-Maghlouth BA, Bahammam MA, Linjawi AI, El-Bialy TH. Corticotomy-assisted orthodontic treatment. A systematic review of the biological basis and clinical effectiveness. Saudi Med J. 2015 Jul;36(7):794-801. doi: 10.15537/smj.2015.7.12437. PMID 26108582
- [Background] Wilcko WM, Wilcko T, Bouquot JE, Ferguson DJ. Rapid orthodontics with alveolar reshaping: two case reports of decrowding. Int J Periodontics Restorative Dent. 2001 Feb;21(1):9-19. PMID 11829041
- [Background] Hassan AH, AlGhamdi AT, Al-Fraidi AA, Al-Hubail A, Hajrassy MK. Unilateral cross bite treated by corticotomy-assisted expansion: two case reports. Head Face Med. 2010 May 19;6:6. doi: 10.1186/1746-160X-6-6. PMID 20482859